CLINICAL TRIAL: NCT04953325
Title: Immunogenicity and Safety of an Inactivated COVID-19 Vaccine for Prevention of COVID-19 in Healthy Population Aged 18 Years and Older
Brief Title: Immunogenicity and Safety of an Inactivated COVID-19 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4004-SD
Record Dates: First submitted 2021-07-05; First posted 2021-07-07 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 180 subjects (including 90 adults aged 18-59 years and 90 elderly aged 60 year and older）will receive two doses of inactivated COVID-19 vaccine on day 0 and day 28
  Interventions: Biological: Inactivated COVID-19 Vaccine
- Control Group (Placebo Comparator): 90 subjects (including 45 adults aged 18-59 years and 45 elderly aged 60 year and older）will receive one dose of 23-valent pneumococcal polysaccharide vaccine on day 0 and one dose of Inactivated Hepatitis A Vaccine on day 28
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: Inactivated Hepatitis A Vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 Vaccine — 600SU inactivated virus in 0·5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Experimental Group
Biological: 23-valent pneumococcal polysaccharide vaccine — 25μg each of the following serotypes/each dose (0.5ml): 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F
  Arms: Control Group
Biological: Inactivated Hepatitis A Vaccine — 500SU inactivated Hepatitis A virus in 1 mL of aluminium hydroxide solution per injection.
  Arms: Control Group

SUMMARY:
This study is a randomized, placebo-controlled and open design, phase 4 clinical trial of an inactivated COVID-19 vaccine (CoronaVac) manufactured by Sinovac Research and Development Co., Ltd. The purpose of this study is to evaluate the immunogenicity and safety of the CoronaVac in healthy population aged 18 years and older.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled and opened, phase 4 clinical trial to evaluate the safety and immunogenicity of an inactivated COVID-19 vaccine(CoronaVac）in healthy population aged 18 years and older . The experimental vaccine is manufactured by Sinovac Research and Development Co.,Ltd. A total of 270 healthy subjects will be enrolled, including 135 adults aged 18-59 years and 135 elderly elderly aged 60 years and older. Subjects in each age group will be divided into two groups in a ratio of 1:1. Subjects in the experimental group will receive two doses of CoronaVac on day 0 and day 28. Subjects in the control group will receive one dose of 23-valent Pneumococcal Polysaccharide Vaccine on day 0 and one dose of Inactivated Hepatitis A Vaccine on day 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy population aged 18 years and above;
* The subjects can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* History of SARS-CoV-2 infection;
* Have received any COVID-19 vaccine;
* Participants with abnormal fasting blood glucose or diabetes;
* History of asthma, history of allergy to the vaccine or vaccine components,or serious adverse reactions to the vaccine, such as urticaria, dyspnea,and angioedema;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, spleenlessness, functional spleenlessness, spleenlessness or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Diseases or factors that are prone to thrombosis or bleeding, such as thrombophlebitis, major surgery/trauma, hereditary thrombotic disorder, sepsis, inflammatory bowel disease, severe varicose veins, May-Thurner syndrome, fibrinolytic activity enhancement disease, history of cardiac stent surgery, allergic purpura, etc.;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Abnormal hematological laboratory test results outside the reference range during previous physical examination within one year: Blood routine indicators (white blood cell count, hemoglobin, platelet count), Coagulation function test (prothrombin time PT, activated partial prothrombin time APTT, fibrinogen FIB, thrombin time TT, international standardized ratio INR, D-dimer), other indicators (blood glucose, platelet factor 4 HIT ELISA, erythrocyte sedimentation rate);
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 3 months;
* History of taking aspirin drugs and other drugs that affect blood coagulation;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of the neutralizing antibody to SARS-CoV-2 | Day 28 after the second dose
  Seroconversion rate of the neutralizing antibody to SARS-CoV-2 at day 28 after the second dose of inactivated COVID-19 vaccine

SECONDARY OUTCOMES:
Seroconversion rate of the neutralizing antibody to SARS-CoV-2 | Day 4, 14, 32,42 and 56 after the first dose
  Seroconversion rate of the neutralizing antibody to SARS-CoV-2 at different points after vaccination
Seropositivity rate of the neutralizing antibody to SARS-CoV-2 | Day 4, 14, 28, 32,42 and 56 after the first dose
  Seropositivity rate of of the neutralizing antibody to SARS-CoV-2 at different points after vaccination
GMT of the neutralizing antibody to SARS-CoV-2 | Day 4, 14, 28, 32,42 and 56 after the first dose
  GMT of of the neutralizing antibody to SARS-CoV-2 at different points after vaccination
GMI of the neutralizing antibody to SARS-CoV-2 | Day 4, 14, 28, 32,42 and 56 after the first dose
  GMT of of the neutralizing antibody to SARS-CoV-2 at different points after vaccination
Geometric mean concentrations of anti-pneumococcal antibody for 23 serotypes (ELISA) | Day 28 after vaccination of 23-valent pneumococcal polysaccharide vaccine
  Geometric mean concentrations of anti-pneumococcal antibody for 23 serotypes (ELISA) at day 28 after vaccination of 23-valent pneumococcal polysaccharide vaccine
Seroconversion rate of anti-pneumococcal antibody for 23 serotypes (ELISA) | Day 28 after vaccination of 23-valent pneumococcal polysaccharide vaccine
  Seroconversion rate of anti-pneumococcal antibody for 23 serotypes (ELISA) at day 28 after vaccination of 23-valent pneumococcal polysaccharide vaccine
Seroconversion rate of the hepatitis A antibody by Electrochemiluminescence | Day 28 after vaccination of Inactivated Hepatitis A Vaccine
  Seroconversion rate of the hepatitis A antibody at day 28 after vaccination of Inactivated Hepatitis A Vaccine
Seropositivity rate of the hepatitis A antibody by Electrochemiluminescence | Day 28 after vaccination of Inactivated Hepatitis A Vaccine
  Seropositivity rate of the hepatitis A antibody at day 28 after vaccination of Inactivated Hepatitis A Vaccine
GMT of the hepatitis A antibody by Electrochemiluminescence | Day 28 after vaccination of Inactivated Hepatitis A Vaccine
  GMT of the hepatitis A antibody at day 28 after vaccination of Inactivated Hepatitis A Vaccine
GMI of the hepatitis A antibody by Electrochemiluminescence | Day 28 after vaccination of Inactivated Hepatitis A Vaccine
  GMI of the hepatitis A antibody at day 28 after vaccination of Inactivated Hepatitis A Vaccine
Occurrence of abnormal changes of laboratory safety examinations | Day 4, 14, 28, 32,42 and 56 after the first dose
  Occurrence of abnormal changes of laboratory safety examinations (Platelet factor 4 HIT, blood sugar, ESR, White blood cell count, hemoglobin, platelet count and Coagulation function index)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (1):
- Rushan City Center for Disease Control and Prevention, Weihai, Shandong, China

REFERENCES:
- [Derived] Xu Q, Lu X, Liu X, Zhao Y, Sun D, Cao Q, Liu H, Yang T, Song Y, Lv J, Xiong P, Li J, Sun J, Xie M, Gao Y, Zhang L. Effect of an inactivated coronavirus disease 2019 vaccine, CoronaVac, on blood coagulation and glucose: a randomized, controlled, open-label phase IV clinical trial. Front Immunol. 2023 May 31;14:1122651. doi: 10.3389/fimmu.2023.1122651. eCollection 2023. PMID 37325662